CLINICAL TRIAL: NCT01692314
Title: Effect of Resistance Training on Microvascular Reactivity, Endothelial Function, Inflammatory Markers, Body Composition, Blood Pressure, Heart Rate and Physical Fitness in Obese Adolescents
Brief Title: Effect of Resistance Training on Microvascular, Hemodynamic and Physical Parameters in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Ingrid Barbara Ferreira Dias, Principal Investigator, Rio de Janeiro State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BIOVASC 2009
Record Dates: First submitted 2012-09-14; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: Endothelial function; Microvascular reactivity; Obesity; Adolescents
MeSH Terms: conditions — Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obese adolescents is being compared to control ones (Experimental): Patients underwent to resistance training, three times a week, during three months.
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training

SUMMARY:
The purpose of this study is to investigate the effect os resistance training on microvascular reactivity, endothelial functions, inflammatory markers, blood pressure, heart rate, body composition and physical fitness in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Tanner pubertal stage of development between three and five
* age between 13 up to 17 years old

Exclusion Criteria:

* presence of chronic diseases (diabetes mellitus, nephropathy and/or hypertension),
* musculoskeletal injury,
* smoking and
* to be in use of any medication.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Microvascular Reactivity | Three months

SECONDARY OUTCOMES:
Endothelial function | Three months

OTHER OUTCOMES:
Hemodynamic parameters | three months
Imflammatory markers | three months
Body composition | three months
Physical fitness | three months

CONTACTS AND LOCATIONS:
Overall Officials: Eliete Bouskela, Phd, Study Director — State University of Rio de Janeiro
Locations (1):
- Laboratory for Clinical and Experimental Research in Vascular Biology (BioVasc), Biomedical Center, State University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil